CLINICAL TRIAL: NCT07137546
Title: Fundus-first Laparoscopic Cholecystectomy in Difficult Gallbladder
Brief Title: Fundus-first Laparoscopic Cholecystectomy
Acronym: FFLC
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Minia University (Other)
Responsible Party: Principal Investigator, Saleh Khairy Saleh MD, Lecturer, Minia University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1131/04/2024
Record Dates: First submitted 2025-08-14; First posted 2025-08-22 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-11

CONDITIONS: Cholecystitis; Acute Cholecystitis; Pericholecystic Abscess
Keywords: Fundus-first laparoscopic cholecystectomy; Conventional laparoscopic cholecystectomy; Bile duct injury; Difficult gallbladder; Critical view of safety
MeSH Terms: conditions — Cholecystitis; Cholecystitis, Acute

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Surgeons are not blinded due to the intervention's nature; data collectors, assessors, and analysts are blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fundus-First Laparoscopic Cholecystectomy ( FFLC) (Experimental): Laparoscopic cholecystectomy starting dissection at the gallbladder fundus, progressing retrograde toward the cystic duct/artery. Critical View of Safety (CVS) confirmed before duct division.
  Interventions: Procedure: Fundus-First Laparoscopic Cholecystectomy ( FFLC)
- Classical Laparoscopic Cholecystectomy (CLC) (Active Comparator): The standard "critical view of safety" technique (anterior-posterior dissection of Calot's triangle first).
  Interventions: Procedure: Classical Laparoscopic Cholecystectomy (CLC)

INTERVENTIONS:
Procedure: Fundus-First Laparoscopic Cholecystectomy ( FFLC) — * Standard 4-port laparoscopic setup
  * Carbon dioxide (CO₂) pneumoperitoneum (12-15 mmHg)
  * Dissection begins at gallbladder fundus
  * Peritoneum incised from infundibulum to fundus along liver bed
  * Gallbladder dissected from fundus toward infundibulum
  * Cystic artery and duct identified and divided last
  * Critical view of safety achieved before vessel division
  Arms: Fundus-First Laparoscopic Cholecystectomy ( FFLC)
Procedure: Classical Laparoscopic Cholecystectomy (CLC) — * Standard 4-port laparoscopic setup
  * Carbon dioxide (CO₂) pneumoperitoneum (12-15 mmHg)
  * Dissection begins at Calot's triangle
  * Critical view of safety achieved first
  * Cystic artery and duct divided before gallbladder bed dissection
  * Gallbladder dissected from liver bed
  Arms: Classical Laparoscopic Cholecystectomy (CLC)

SUMMARY:
Bile duct injury (BDI) remains the most feared complication of laparoscopic cholecystectomy, particularly in difficult gallbladder cases. The fundus-first technique has emerged as a potentially safer alternative to classical laparoscopic cholecystectomy for challenging cases. This single-center, prospective, randomized controlled trial compared the efficacy and safety of fundus-first laparoscopic cholecystectomy (FF-LC) versus classical laparoscopic cholecystectomy (C-LC) in 174 patients with difficult gallbladder characteristics. The primary outcome was bile duct injury rate. Secondary outcomes included conversion to open surgery, operative parameters, and postoperative complications.

DETAILED DESCRIPTION:
Bile duct injury (BDI) rates remain 0.3-1.5% in difficult gallbladders. FFLC avoids early dissection near critical structures, potentially lowering BDI risk.

This randomized controlled trial aims to compare the safety and efficacy of fundus-first (FF) versus classical (Calot-first) laparoscopic cholecystectomy techniques in patients with difficult gallbladders. The study will evaluate perioperative outcomes, conversion rates, complications, and operative time between the two surgical approaches. Based on recent evidence suggesting an improved safety profile with the fundus-first technique, we hypothesize that the FF approach will demonstrate reduced bile duct injury rates and improved surgical outcomes in difficult cases.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-80 years
* Symptomatic cholelithiasis or cholecystitis requiring laparoscopic cholecystectomy (elective or emergency)
* Difficult gallbladder characteristics: Acute cholecystitis (Tokyo Guidelines 2018 Grade II/III), wall thickness >4 mm on US, pericholecystic fluid, impacted stone in Hartmann's pouch/cystic duct, previous upper abdominal surgery, BMI >30 kg/m², ≥3 previous cholecystitis episodes, contracted gallbladder, Mirizzi syndrome Type I/II, empyema, severe pericholecystic adhesions on imaging, suspected anatomical variations
* The American Society of Anesthesiologists (ASA) physical status I-III
* Suitable for laparoscopic approach
* Informed consent

Exclusion Criteria:

* Suspected gallbladder malignancy
* Choledocholithiasis requiring endoscopic intervention
* Mirizzi syndrome Grade III-IV
* Gallbladder perforation with generalized peritonitis
* Pregnancy or lactation
* Contraindications to laparoscopy (severe cardiopulmonary disease, coagulopathy)
* Previous biliary or hepatic surgery
* Cirrhosis with portal hypertension
* Active coagulopathy
* Patient refusal

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 174 (Actual)
Dates: Start 2024-05-01 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Bile Duct Injury Rate | Intraoperative to 30 days postoperative
  Incidence of bile duct injury, confirmed by intraoperative cholangiography, direct visualization, or postoperative imaging.

SECONDARY OUTCOMES:
Conversion to Open Surgery Rate | Intraoperative
  Rate of conversion from laparoscopic to open procedure due to dense adhesions, bleeding, unclear anatomy, or suspected BDI.
Operative Time | Intraoperative
  Total time from skin incision to closure (minutes).
Time to Achieve Critical View of Safety (CVS) | Intraoperative
  Time from incision to CVS achievement (minutes).
CVS Achievement Rate | Intraoperative
  Proportion of cases where CVS was achieved.
Estimated Blood Loss | Intraoperative
  Intraoperative blood loss (mL).
Intraoperative Cholangiography Rate | Intraoperative
  Proportion requiring cholangiography for unclear anatomy or suspected stones.
Gallbladder Perforation Rate | Intraoperative
  Incidence of intraoperative gallbladder perforation.

OTHER OUTCOMES:
Intraoperative Complications Rate | Intraoperative
  Overall intraoperative complications (e.g., bleeding, perforation, injury).
Postoperative Complications | Up to 30 days postoperative
  Rate of complications requiring treatment or intervention.
Major Postoperative Complications | Up to 30 days postoperative
  Rate of complications requiring surgical intervention under anesthesia.
Length of Hospital Stay | Postoperative
  Days from surgery to discharge .
Readmission Rate Within 30 Days | 30 days postoperative
  Proportion readmitted for complications.
Time to Return to Normal Activity | Up to 30 days postoperative
  Days to resume normal activities

CONTACTS AND LOCATIONS:
Overall Officials: Saleh K Saleh, MD, Principal Investigator — Minia University
Locations (1):
- Liver and GIT hospital / Minia university, Minya, Minya Governorate, Egypt